CLINICAL TRIAL: NCT00307801
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled, 7 Cycle Duration (196 Days), Phase 3 Study of Oral Estradiol Valerate/Dienogest Tablets for the Treatment of Dysfunctional Uterine Bleeding.
Brief Title: Efficacy and Safety Study for the Treatment of Dysfunctional Uterine Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91470; 2005-004340-32 (EudraCT Number); 308961 (Other: Company internal)
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Metrorrhagia
Keywords: Dysfunctional uterine bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Estradiol; dienogest

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estradiol valerate/Dienogest (Natazia, Qlaira, BAY86-5027) (Experimental): A blister consists of 28 tablets taken orally once a day for 28 days (one cycle): 2 days of 3 mg estradiol valerate (EV); 5 days of 2 mg EV + 2 mg dienogest (DNG); 17 days of 2 mg EV + 3 mg DNG; 2 days of 1 mg EV; 2 days of placebo.
  Interventions: Drug: Estradiol valerate/Dienogest (Natazia, Qlaira, BAY86-5027)
- Placebo (Placebo Comparator): Matching placebo to be taken orally daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol valerate/Dienogest (Natazia, Qlaira, BAY86-5027) — 1 pill per day taken orally over 7 cycles of 28 pills per cycle
  Arms: Estradiol valerate/Dienogest (Natazia, Qlaira, BAY86-5027)
Drug: Placebo — 1 pill per day taken orally over 7 cycles of 28 pills per cycle
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the study drug is safe and effective in the treatment of dysfunctional uterine bleeding.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer HealthCare AG, Germany. Bayer HealthCare AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older
* And with a diagnosis of dysfunctional uterine bleeding without organic pathology
* And with at least one of the following symptoms: prolonged, frequent or excessive bleeding.

Exclusion Criteria:

* The use of steroidal oral contraceptives, or any drug that could alter oral contraception metabolism will be prohibited during the study.
* Women with a history of endometrial ablation or dilatation and curettage within 2 months prior to study start will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2006-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (36):
- Australia (2):
  - Private Practice Dr. Ian Fraser, Ashfield, New South Wales
  - King Edward Memorial Hospital, Subiaco, Western Australia
- Czechia (4):
  - Gynekologicka ambulance Vanda Horejsi, MD, České Budějovice
  - Center for Clinical& Basic Research, Pardubice
  - Gynekologicko-poradnicka ambulance Dr. Hlavackova, Písek
  - Lekarsky dum Praha 7 a.s.Gynekologicka ambulance Dr. Jenicek, Prague
- Finland (4):
  - Adenova Lääkärikeskus Oy, Espoo
  - Terveystalo Lahti, Lahti
  - Koskiklinikka, Tampere
  - Ylioppilaiden terveydenhoitosäätiö, Turku, Turku
- Germany (5):
  - Praxis Hr. Dr. U. Kohoutek, Karlsruhe, Baden-Wurttemberg
  - Praxis Hr. Dr. S. Schönian, Rheinstetten, Baden-Wurttemberg
  - Praxis Hr. Dr. K. Greven, Hanover, Lower Saxony
  - ClinPharm International GmbH, Dresden, Saxony
  - emovis GmbH, Berlin, State of Berlin
- Hungary (3):
  - University of Semmelweis, Budapest
  - Selya Janos Hospital, Komárom
  - Borsod-Abauj-Zemplen County Hospital, Miskolc
- Netherlands (3):
  - Medisch Spectrum Twente, Locatie Ariensplein, Enschede
  - PreCare Trial & Recruitment, Geleen
  - Menox BV, Nijmegen
- Poland (5):
  - Poliklinika Ginekologiczna- Poloznicza, Bialystok
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - SPSK nr 1, Lublin
  - Szpital Kliniczny nr 3, Poznan
  - CSK MSWiA, Warsaw
- Sweden (3):
  - Skånes Universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Ukraine (4):
  - Dept. of obstetrics and gynaecology, Kiev
  - Instr. of Pediatrics, Obstetrics & Gynecology, Kiev
  - Kyiv Medical Academy of Postdyploma Education, Kiev
  - Lviv Regional Center Perinatal Center, Lviv
- United Kingdom (3):
  - Bridge House Medical Centre, Cheadle, Cheshire
  - Luton & Dunstable Hospital, Luton
  - MeDiNova Research, Northwood

REFERENCES:
- [Result] Fraser IS, Jensen J, Schaefers M, Mellinger U, Parke S, Serrani M. Normalization of blood loss in women with heavy menstrual bleeding treated with an oral contraceptive containing estradiol valerate/dienogest. Contraception. 2012 Aug;86(2):96-101. doi: 10.1016/j.contraception.2011.11.011. Epub 2012 Jan 10. PMID 22240178
- [Result] Fraser IS, Parke S, Mellinger U, Machlitt A, Serrani M, Jensen J. Effective treatment of heavy and/or prolonged menstrual bleeding without organic cause: pooled analysis of two multinational, randomised, double-blind, placebo-controlled trials of oestradiol valerate and dienogest. Eur J Contracept Reprod Health Care. 2011 Aug;16(4):258-69. doi: 10.3109/13625187.2011.591456. PMID 21774563
- [Result] Fraser IS, Romer T, Parke S, Zeun S, Mellinger U, Machlitt A, Jensen JT. Effective treatment of heavy and/or prolonged menstrual bleeding with an oral contraceptive containing estradiol valerate and dienogest: a randomized, double-blind Phase III trial. Hum Reprod. 2011 Oct;26(10):2698-708. doi: 10.1093/humrep/der224. Epub 2011 Jul 21. PMID 21784734
- [Result] Wasiak R, Filonenko A, Vanness DJ, Wittrup-Jensen KU, Stull DE, Siak S, Fraser I. Impact of estradiol-valerate/dienogest on work productivity and activities of daily living in European and Australian women with heavy menstrual bleeding. Int J Womens Health. 2012;4:271-8. doi: 10.2147/IJWH.S31740. Epub 2012 Jul 12. PMID 22927764
- [Result] Fraser IS, Zeun S, Parke S, Wilke B, Junge W, Serrani M. Improving the objective quality of large-scale clinical trials for women with heavy menstrual bleeding: experience from 2 multi-center, randomized trials. Reprod Sci. 2013 Jul;20(7):745-54. doi: 10.1177/1933719113477492. Epub 2013 Feb 25. PMID 23439617
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of first subject first visit was 16 Feb 2006. The date of last visit last subject was 27 May 2008.
Pre-assignment Details: A total of 575 subjects were screened for inclusion into the study. 344 failed screening. The remaining 231 were randomized.
Period: Overall Study
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Started | 149 | 82
Subjects Received Treatment | 145 | 81
Cycle 1, Visit 5, Baseline | 145 | 81
Cycle 3, Visit 7, Treatment Day 84 | 130 | 71
Cycle 7, Treatment Day 196 | 141 (Includes subjects that prematurely discontinued the study and may not be counted in earlier visits.) | 77 (Includes subjects that prematurely discontinued the study and may not be counted in earlier visits.)
Completed | 117 | 65
Not Completed | 32 | 17
Not completed — Adverse Event | 12 | 4
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Non-compliance, not taken all tablets | 1 | 2
Not completed — Adverse event (AE)/Withdrawal of consent | 2 | 0
Not completed — Decreased Libido (AE at discontinuation) | 0 | 1
Not completed — Wrong Randomization | 1 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up, moved abroad | 1 | 1
Not completed — Frustration with e-diary | 1 | 0
Not completed — Protocol Violation | 3 | 2
Not completed — No reason specified | 2 | 0
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo | Total
Number analyzed (Participants) | 149 | 82 | 231
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (6.6) | 38.5 (7.5) | 39.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 82 | 231
  Male | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Body mass index was calculated with body weight and height measured at screening (BMI = body weight in kg/ body height in m^2)
  kg/m² | 24.5 (3.5) | 25.7 (3.0) | 24.9 (3.4)
excessive bleeding [Number; unit: participants] — Excessive bleeding: 2 or more bleeding episodes each with blood loss volume of 80 mL or more in a 90-day period, as assessed by the alkaline hematin method.
  participants | 136 | 76 | 212
prolonged bleeding [Number; unit: participants] — Prolonged bleeding: 2 or more bleeding episodes, each lasting 8 or more days.
  participants | 20 | 10 | 30
frequent bleeding [Number; unit: participants] — Frequent bleeding: greater than 5 bleeding episodes, with a minimum of 20 bleeding days overall.
  participants | 0 | 0 | 0
prolonged and frequent bleeding [Number; unit: participants] — Prolonged bleeding: 2 or more bleeding episodes, each lasting 8 or more days.Frequent bleeding: greater than 5 bleeding episodes, with a minimum of 20 bleeding days overall.
  participants | 0 | 0 | 0
prolonged and excessive bleeding [Number; unit: participants] — Prolonged bleeding: 2 or more bleeding episodes, each lasting 8 or more days. Excessive bleeding: 2 or more bleeding episodes each with blood loss volume of 80 mL or more in a 90-day period, as assessed by the alkaline hematin method.
  participants | 15 | 9 | 24
frequent and excessive bleeding [Number; unit: participants] — Excessive bleeding: 2 or more bleeding episodes each with blood loss volume of 80 mL or more in a 90-day period, as assessed by the alkaline hematin method. Frequent bleeding: greater than 5 bleeding episodes, with a minimum of 20 bleeding days overall.
  participants | 0 | 0 | 0
prolonged, frequent and excessive bleeding [Number; unit: participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With no Dysfunctional Uterine Bleeding (DUB) Symptoms
Description: At least 6, up to 8 criteria to be met in complete response during 90-day period: no bleeding episodes(BE) >7 days, no >4 BE, no BE with blood loss (menstrual blood loss, MBL) ≥80 mL, no >1 BE increase from baseline, no increase from baseline in individual patient's total number of bleeding days and total number of bleeding days not >24 days. Additionally, for subjects included with prolonged bleeding: decrease between maximum duration during run-in and efficacy ≥2 days excessive bleeding: MBL associated with each episode decreased by ≥50% from average of qualifying episodes during run-in.
Time Frame: Efficacy phase was defined as a 90-day period under treatment. For patients who completed up to day 6 of treatment cycle 7, the efficacy phase started on the first day of treatment cycle 4, and continued through day 6 of treatment cycle 7
Population: Intent-To-Treat (ITT): all randomized subjects with ≥1 of the DUB symptoms in 90-day run-in phase: Prolonged bleeding: ≥2 bleeding episodes, each lasting ≥8 days Frequent bleeding: >5 bleeding episodes, with minimum of 20 bleeding days overall. Excessive bleeding: ≥2 bleeding episodes each with blood loss volume (=MBL) of ≥80 mL
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 149 | 82
Proportion of participants | 0.295 | 0.012
Statistical Analysis 1: Comparison: Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) vs Placebo; Test type: Superiority or Other; p < 0.0001, inverting 2 one-sided tests

2. Secondary Outcome: Proportion of Participants Cured From Prolonged Bleeding
Description: Prolonged bleeding: 2 or more bleeding episodes, each lasting 8 or more days. Cure from prolonged bleeding: no bleeding episodes lasting more than 7 days and the decrease between maximum duration during run-in and maximum duration during the efficacy phase was at least 2 days.
Time Frame: as for outcome 1
Population: The ITT population consisted of all randomized subjects with prolonged bleeding: 2 or more bleeding episodes, each lasting 8 or more days
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 20 | 10
Proportion of participants | 0.350 | 0.100

3. Secondary Outcome: Proportion of Participants Cured From Excessive Bleeding
Description: Excessive bleeding:>=2 bleeding episodes each with blood loss volume (MBL) of >=80 mL in 90-day period, assessed by alkaline hematin method. This spectrophotometrical method measures hemoglobin (Hb) in fixed amount of alkaline solution, taken from pool of solution in which materials (used sanitary protection) to be tested have been macerated for Hb extraction. Cure from excessive bleeding: MBL in each episode <80 mL + blood loss volume associated with each bleeding episode is decrease of ≥50% from average of qualifying bleeding episodes (with blood loss volume ≥80 mL per episode during run-in)
Time Frame: as for outcome 1
Population: The ITT population consisted of all randomized subjects who enrolled with excessive bleeding: 2 or more bleeding episodes each with blood loss volume of 80 mL or more in a 90-day run-in period, as assessed by the alkaline hematin method
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 136 | 76
Proportion of participants | 0.441 | 0.013

4. Secondary Outcome: Proportion of Participants Cured From Frequent Bleeding
Description: Frequent bleeding: greater than 5 bleeding episodes, with a minimum of 20 bleeding days overall. Cure from frequent bleeding: no more than 4 bleeding episodes and the total number of bleeding days did not exceed 24 days and no increase from baseline in an individual patient's total number of bleeding days occurred
Time Frame: as for outcome 1
Population: The ITT population consisted of all randomized subjects who enrolled with frequent bleeding: greater than 5 bleeding episodes, with a minimum of 20 bleeding days overall
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Proportion of Participants With Improvement in the Investigator's Global Assessment Scale at Treatment Day 84
Description: According to the investigator's global assessment scale "improved" was defined as being classified as 'very much improved', 'much improved', or 'improved' and "not improved" was defined as being classified as 'no change', 'worse', 'much worse', 'very much worse', or 'not assessed'. Central laboratory data, physical examination, e-diary data, and patient interview were used as sources for the assessment at day 84 compared with admission to study data.
Time Frame: From baseline (visit 5, day 1) up to treatment day 84
Population: ITT, all participants with assessment at day 84 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 130 | 71
Proportion of participants | 0.838 | 0.394

6. Secondary Outcome: Proportion of Participants With Improvement in the Investigator's Global Assessment Scale at Treatment Day 196
Description: According to the investigator's global assessment scale "improved" was defined as being classified as 'very much improved', 'much improved', or 'improved' and "not improved" was defined as being classified as 'no change', 'worse', 'much worse', 'very much worse', or 'not assessed'. Central laboratory data, physical examination, e-diary data, and patient interview were used as sources for the assessment at day 196 compared with admission to study data.
Time Frame: From baseline (visit 5, day 1) up to treatment day 196
Population: ITT, all participants with assessment at day 196 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 144 | 81
Proportion of participants | 0.847 | 0.395

7. Secondary Outcome: Proportion of Participants With Improvement in the Patient's Overall Assessment Scale at Treatment Day 84
Description: According to the patient's global assessment scale "improved" was defined as being classified as 'very much improved', 'much improved', or 'improved' and "not improved" was defined as being classified as 'no change', 'worse', 'much worse', 'very much worse', or 'not assessed'. Patients assessed the overall improvement at day 84 compared with admission to the study condition.
Time Frame: From baseline (visit 5, day 1) up to treatment day 84
Population: ITT, all participants with assessment at day 84 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 127 | 68
Proportion of participants | 0.724 | 0.529

8. Secondary Outcome: Proportion of Participants With Improvement in the Patient's Overall Assessment Scale at Treatment Day 196
Description: According to the patient´s global assessment scale "improved" was defined as being classified as 'very much improved', 'much improved', or 'improved' and "not improved" was defined as being classified as 'no change', 'worse', 'much worse', 'very much worse', or 'not assessed'. Patients assessed the overall improvement at day 196 compared with admission to the study condition.
Time Frame: From baseline (visit 5, day 1) up to treatment day 196
Population: ITT, all participants with assessment at day 196 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 136 | 71
Proportion of participants | 0.779 | 0.451

9. Secondary Outcome: Change From Baseline in Blood Loss Volume for All Participants to the Reference Period of 90 Days Under Treatment
Description: Menstrual blood loss volume as assessed by the alkaline hematin method for the 90 days before treatment (baseline) and for 90 days under treatment. This spectrophotometrical method measures hemoglobin (Hb) in fixed amount of alkaline solution, taken from pool of solution in which materials (used sanitary protection) to be tested have been macerated for Hb extraction. A negative value indicates a reduction in blood loss after treatment.
Time Frame: Baseline and reference period of 90 days under treatment. For patients who completed up to day 6 of treatment cycle 7, the efficacy phase started on the first day of treatment cycle 4, and continued through day 6 of treatment cycle 7
Population: ITT, all participants with assessments at baseline and efficacy phase for this outcome measure
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 108 | 60
ml | -458.4 (409.6) | -93.2 (268.0)

10. Secondary Outcome: Menstrual Blood Loss Volume for All Participants at Cycle 1
Description: Menstrual blood loss volume as assessed by the alkaline hematin method after patients were on treatment for one cycle. This spectrophotometrical method measures hemoglobin (Hb) in fixed amount of alkaline solution, taken from pool of solution in which materials (used sanitary protection) to be tested have been macerated for Hb extraction.
Time Frame: Cycle 1 = 28 days (one cycle)
Population: ITT, all participants with assessments for this outcome measure
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 144 | 81
ml | 175.6 (188.3) | 194.3 (171.1)

11. Secondary Outcome: Menstrual Blood Loss Volume for All Participants at Cycle 3
Description: Menstrual blood loss volume as assessed by the alkaline hematin method after patients were on treatment for 3 cycles. This spectrophotometrical method measures hemoglobin (Hb) in fixed amount of alkaline solution, taken from pool of solution in which materials (used sanitary protection) to be tested have been macerated for Hb extraction.
Time Frame: Cycle 3 = 28 days (one cycle)
Population: ITT, all participants with assessments for this outcome measure
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 136 | 73
ml | 68.3 (111.6) | 195.1 (161.8)

12. Secondary Outcome: Menstrual Blood Loss Volume for All Participants at Cycle 7
Description: Menstrual blood loss volume as assessed by the alkaline hematin method after patients were on treatment for 7 cycles. This spectrophotometrical method measures hemoglobin (Hb) in fixed amount of alkaline solution, taken from pool of solution in which materials (used sanitary protection) to be tested have been macerated for Hb extraction.
Time Frame: Cycle 7 = 28 days (one cycle)
Population: ITT, all participants with assessments for this outcome measure
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 111 | 63
ml | 44.6 (70.9) | 167.2 (112.2)

13. Secondary Outcome: Change From Baseline in Blood Loss Volume for Participants With Excessive Bleeding to the Reference Period of 90 Days Under Treatment.
Description: Blood loss volume as assessed by the alkaline hematin method for participants with excessive bleeding (2 or more bleeding episodes each with blood loss volume of 80 ml or more during the run-in phase) for the 90 days before treatment (ie, run-in phase) and for the 90 days under treatment. A negative value indicates a reduction in blood loss while under treatment compared to before treatment.
Time Frame: as for outcome 9
Population: ITT consisted of all randomized subjects enrolled with excessive bleeding. This spectrophotometrical method measures hemoglobin (Hb) in fixed amount of alkaline solution, taken from pool of solution in which materials (used sanitary protection) to be tested have been macerated for Hb extraction.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 102 | 59
ml | -480.6 (410.6) | -94.2 (270.2)

14. Secondary Outcome: Menstrual Blood Loss Volume for Participants With Excessive Bleeding at Cycle 1.
Description: Blood loss volume as assessed by the alkaline hematin method for participants with excessive bleeding (2 or more bleeding episodes each with blood loss volume of 80 ml or more during the run-in phase) after participants were on treatment for one cycle. This spectrophotometrical method measures hemoglobin (Hb) in fixed amount of alkaline solution, taken from pool of solution in which materials (used sanitary protection) to be tested have been macerated for Hb extraction.
Time Frame: Cycle 1 = 28 days (one cycle)
Population: ITT consisted of all randomized subjects enrolled with excessive bleeding: 2 or more bleeding episodes each with blood loss volume of 80 mL or more, as assessed by the alkaline hematin method.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 133 | 75
ml | 207.8 (186.1) | 238.9 (196.0)

15. Secondary Outcome: Menstrual Blood Loss Volume for Participants With Excessive Bleeding at Cycle 3.
Description: Blood loss volume as assessed by the alkaline hematin method for participants with excessive bleeding (2 or more bleeding episodes each with blood loss volume of 80 ml or more during the run-in phase) after participants were on treatment for 3 cycles. This spectrophotometrical method measures hemoglobin (Hb) in fixed amount of alkaline solution, taken from pool of solution in which materials (used sanitary protection) to be tested have been macerated for Hb extraction.
Time Frame: Cycle 3 = 28 days (one cycle)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 126 | 68
ml | 72.1 (115.0) | 188.4 (150.1)

16. Secondary Outcome: Menstrual Blood Loss Volume for Participants With Excessive Bleeding at Cycle 7.
Description: Blood loss volume as assessed by the alkaline hematin method for participants with excessive bleeding (2 or more bleeding episodes each with blood loss volume of 80 ml or more during the run-in phase) after participants were on treatment for 7 cycles. This spectrophotometrical method measures hemoglobin (Hb) in fixed amount of alkaline solution, taken from pool of solution in which materials (used sanitary protection) to be tested have been macerated for Hb extraction.
Time Frame: Cycle 7 = 28 days (one cycle)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 104 | 60
ml | 46.7 (72.7) | 168.6 (112.6)

17. Secondary Outcome: Change From Baseline in Number of Bleeding Episodes to the Reference Period of 90 Days Under Treatment
Description: A bleeding episode is characterized by the following: • Bleeding for at least 2 days • Bleeding days can be separated by no more than 1 bleeding-free day • An episode stops with 2 consecutive bleeding-free days. The number of episodes was determined for the 90 days before treatment and for the 90 days under treatment. negative value indicates a reduction from baseline in the number of episodes while under treatment.
Time Frame: as for outcome 9
Population: ITT, all participants with assessments at baseline and efficacy phase for this outcome measure
Measure: Mean (Standard Deviation); unit: Bleeding episodes
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 108 | 60
Bleeding episodes | -0.35 (1.09) | -0.38 (0.74)

18. Secondary Outcome: Change From Baseline in Number of Bleeding Days to the Reference Period of 90 Days Under Treatment
Description: A bleeding day is a day on which sanitary protection is required. The number of bleeding days was determined for the 90 days before treatment (baseline) and for 90 days while under treatment. A negative value indicates a reduction in the number of bleeding days while under treatment compared to baseline.
Time Frame: as for outcome 9
Population: ITT, all participants with assessments at baseline and efficacy phase for this outcome measure
Measure: Mean (Standard Deviation); unit: Bleeding days
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 108 | 60
Bleeding days | -5.13 (9.72) | -3.08 (7.88)

19. Secondary Outcome: Change From Baseline in Number of Sanitary Protection Used at 90 Days of Treatment
Description: The number of total sanitary protection items used during the 90 days before treatment (baseline) and those used during the 90 days while under treatment was determined. A negative value indicates a reduction in the number of sanitary protection items used while under treatment compared to baseline.
Time Frame: as for outcome 9
Population: ITT, all participants with assessments for baseline and efficacy phase for this outcome measure
Measure: Mean (Standard Deviation); unit: Sanitary protection products
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 108 | 60
Sanitary protection products | -38.4 (30.0) | -16.5 (32.2)

20. Secondary Outcome: Change From Baseline in Hemoglobin Concentration at Treatment Day 84
Description: Hemoglobin was measured before treatment and after 84 days under treatment. A positive value indicates an increase in hemoglobin from baseline at treatment day 84.
Time Frame: Baseline (visit 5) and treatment day 84
Population: ITT, all participants with assessments at baseline and day 84 for this outcome measure
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 129 | 70
g/dL | 0.36 (0.90) | 0.12 (0.91)

21. Secondary Outcome: Change From Baseline in Hemoglobin Concentration at Treatment Day 196
Description: Hemoglobin was measured before treatment and after 196 days under treatment. A positive value indicates an increase in hemoglobin from baseline at treatment day 196.
Time Frame: Baseline (visit 5) and treatment day 196
Population: ITT, all participants with assessments at baseline and day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 137 | 76
g/dL | 0.70 (1.19) | 0.06 (0.90)

22. Secondary Outcome: Change From Baseline in Hematocrit at Treatment Day 196.
Description: Hematocrit was measured before treatment and after 196 days under treatment. A positive value indicates an increase in hematocrit from baseline at treatment day 196.
Time Frame: Baseline (visit 5) and treatment day 196
Population: ITT, all participants with assessments at baseline and day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 136 | 76
ng/mL | 1.63 (4.25) | 0.08 (3.12)

23. Secondary Outcome: Change From Baseline in Ferritin Concentration at Treatment Day 84
Description: Ferritin was measured before treatment and after 84 days under treatment. A positive value indicates an increase in ferritin from baseline at treatment day 84.
Time Frame: Baseline (visit 5, day 1) and treatment day 84
Population: ITT, all participants with assessments at baseline and treatment day 84 for this outcome measure
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 130 | 71
ng/mL | 2.8 (10.7) | 0.0 (13.7)

24. Secondary Outcome: Change From Baseline in Ferritin Concentration at Treatment Day 196
Description: Ferritin was measured before treatment and after 196 days under treatment. A positive value indicates an increase in ferritin from baseline at treatment day 196.
Time Frame: Baseline (visit 5, day 1) and treatment day 196
Population: ITT, all participants with assessments at baseline and treatment day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 137 | 77
ng/mL | 8.6 (18.5) | 0.5 (12.4)

25. Secondary Outcome: Change From Baseline in Psychological General Well-Being Index (PGWBI) Score at Treatment Day 84.
Description: The PGWBI questionnaire consisted of 22 questions that were answered using a 6-grade Likert scale. The minimum overall score was 22 and the maximum 132. The higher the score, the better the well-being of the patient. The observation phase was the last 4 weeks. The following 6 dimensions were derived from the questionnaire: anxiety, depressed mood, positive well-being, self-control, health, and vitality and the highest possible scores were 30, 18, 24, 18, 18, and 24, respectively.
Time Frame: Baseline (visit 5, day 1) and treatment day 84
Population: ITT, all participants with assessments at baseline and treatment day 84 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 121 | 65
Scores on a scale | -1.2 (13.6) | 2.2 (12.1)

26. Secondary Outcome: Change From Baseline in Psychological General Well-Being Index (PGWBI) Score at Treatment Day 196.
Description: as for outcome 25
Time Frame: Baseline (visit 5, day 1) and treatment day 196
Population: ITT, all participants with assessments at baseline and treatment day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 127 | 68
Scores on a scale | -2.3 (13.6) | 4.6 (11.0)

27. Secondary Outcome: Change From Baseline in McCoy Female Sexuality Questionnaire (MFSQ) Score at Treatment Day 84
Description: The MFSQ was designed to measure aspects of female sexuality and asked about the patients´sexual experience during the last 4 weeks. Higher scores represent higher, more complete, or better integrated levels of female sexual function. Minimum and maximum values are 19 and 133.
Time Frame: Baseline (visit 5, day 1) and treatment day 84
Population: ITT, all participants with assessments at baseline and treatment day 84 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 60 | 25
Scores on a scale | -1.2 (9.1) | 0.4 (8.2)

28. Secondary Outcome: Change From Baseline in McCoy Female Sexuality Questionnaire (MFSQ) Score at Treatment Day 196
Description: as for outcome 27
Time Frame: Baseline (visit 5, day 1) and treatment day 196
Population: ITT, all participants with assessments at baseline and treatment day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 67 | 28
Scores on a scale | -4.9 (11.8) | -2.4 (12.3)

29. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensional (EQ-5D) Score at Treatment Day 84
Description: The health state classification of the EQ-5D comprises 5 questions addressing mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Patients were asked to indicate their current health state by ticking the most appropriate of 3 statements about each of the questions (ie, no problems, some problems, extreme problems). The best possible answers were (1,1,1,1,1), which equals a valuation score of 1.0. The worst possible answers were (3,3,3,3,3), which equals a score of .594.
Time Frame: Baseline (visit 5, day 1) and treatment day 84
Population: ITT, all participants with assessments at baseline and treatment day 84 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 123 | 66
Scores on a scale | -0.0041 (0.1209) | 0.0082 (0.1400)

30. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensional (EQ-5D) Score at Treatment Day 196
Description: as for outcome 29
Time Frame: Baseline (visit 5, day 1) and treatment day 196
Population: ITT, all participants with assessments at baseline and treatment day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 133 | 70
Scores on a scale | -0.0191 (0.1612) | 0.0116 (0.1642)

31. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) of the EQ-5D Score at Treatment Day 84.
Description: The visual analogue scale (ie, "thermometer") had endpoints of 100 (best imaginable health state) at the top, and 0 (worst imaginable health state) at the bottom. Patients rated their current health state by drawing a line from the box marked "your own health state today" to the appropriate point on the thermometer scale.
Time Frame: Baseline (visit 5, day 1) and treatment day 84
Population: ITT, all participants with assessments at baseline and treatment day 84 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 123 | 66
Scores on a scale | -1.63 (13.31) | 0.62 (12.95)

32. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) of the EQ-5D Score at Treatment Day 196.
Description: as for outcome 31
Time Frame: Baseline (visit 5, day 1) and treatment day 196
Population: ITT, all participants with assessments at baseline and treatment day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 131 | 68
Scores on a scale | -3.00 (15.02) | 2.69 (13.68)

33. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Change in the Employment Status） at Treatment Day 84.
Description: The patient was asked if there was any change in her employment status in the last 12 weeks and was asked to specify the number of hours per week. The proportion of participants with such changes are displayed.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 126 | 66
Proportion of participants | 0.095 | 0.152

34. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Change in the Employment Status） at Treatment Day 196.
Description: as for outcome 33
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 133 | 69
Proportion of participants | 0.098 | 0.087

35. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Days Missed From Work） at Treatment Day 84
Description: The patient was asked how many days and hours she missed from work during the past 12 weeks because of her problems associated with her DUB, not including the time missed to participate in this study.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 96 | 52
days | 0.14 (0.776) | 0.27 (1.140)

36. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Days Missed From Work） at Treatment Day 196
Description: as for outcome 35
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 112 | 52
days | 0.13 (0.667) | 0.52 (1.904)

37. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Productivity While Working） at Treatment Day 84.
Description: The patient was asked to rate on a scale of 0 to 10, how much her DUB affected her productivity while she was working during the past 12 weeks, where 0 represented that her DUB had no effect on her work and 10 represented that her DUB completely prevented her from working.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 114 | 61
Scores on a scale | 2.0 (1.71) | 3.1 (2.49)

38. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Productivity While Working） at Treatment Day 196.
Description: as for outcome 37
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 125 | 60
Scores on a scale | 1.8 (1.77) | 3.1 (2.51)

39. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Regular Daily Activities） at Treatment Day 84
Description: The patient was asked to rate on a scale of 0 to 10, how much her DUB affected her ability to do her regular daily activities, other than work at a job, during the past 12 weeks, where 0 represented that her DUB had no effect on her daily activities and 10 represented that her DUB completely prevented her from doing her daily activities.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 118 | 63
Scores on a scale | 2.1 (1.75) | 3.2 (2.39)

40. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Regular Daily Activities） at Treatment Day 196.
Description: as for outcome 39
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 126 | 61
Scores on a scale | 2.0 (1.79) | 3.2 (2.46)

41. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Unscheduled Outpatient Visit at Hospital） at Treatment Day 84
Description: The patient was asked if she had any unscheduled outpatient visits to a hospital because of her DUB during the past 12 weeks, not including visits that were due to her participation in this study. She was also asked to indicate the number of visits. The proportion of participants with any unscheduled outpatient visits are displayed.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 121 | 66
Proportion of participants | 0.008 | 0.0

42. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Unscheduled Outpatient Visit at Hospital） at Treatment Day 196
Description: as for outcome 41
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 131 | 68
Proportion of participants | 0.008 | 0.0

43. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Unscheduled Outpatient Visit to Physician） at Treatment Day 84
Description: The patient was asked if she had any unscheduled outpatient visits to a physician (non-hospital medical care) because of her DUB during the past 12 weeks, not including visits that were due to her participation in this study. She was also asked to indicate the number of visits. The proportion of participants with such visits are displayed.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 121 | 65
Proportion of participants | 0.058 | 0.031

44. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Unscheduled Outpatient Visit to Physician） at Treatment Day 196
Description: as for outcome 43
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 130 | 66
Proportion of participants | 0.031 | 0.015

45. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Additional Unscheduled Procedures） at Treatment Day 84
Description: The patient was asked if she had any unscheduled procedures (eg, laparoscopy, laboratory tests, ultrasound) because of her DUB during the past 12 weeks. The proportion of participants with such procedures are displayed.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 120 | 65
Proportion of participants | 0.0 | 0.0

46. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Additional Unscheduled Procedures） at Treatment Day 196
Description: as for outcome 45
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 128 | 61
Proportion of participants | 0.0 | 0.0

47. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Received Ambulatory Services） at Treatment Day 84
Description: The patient was asked if she received ambulatory services (eg, home help, child care) because of her DUB during the past 12 weeks, and if yes, how many hours per week. The proportion of participants with such services are displayed.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 117 | 65
Proportion of participants | 0.0 | 0.0

48. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Received Ambulatory Services） at Treatment Day 196
Description: as for outcome 47
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 130 | 63
Proportion of participants | 0.0 | 0.0

49. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （no Out-of-pocket Expenses） at Treatment Day 84
Description: The patient was asked to specify her out-of pocket expenses because of her DUB during the past 12 weeks, including over-the-counter medication (the name of the medication, the number of packages, and the cost per package), co-payments due to prescribed medication, and costs to travel to and from medical appointments. The proportion of participants with no out-of pocket expenses are displayed.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 124 | 67
Proportion of participants | 0.855 | 0.881

50. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （no Out-of-pocket Expenses） at Treatment Day 196
Description: as for outcome 49
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 137 | 66
Proportion of participants | 0.920 | 0.879

51. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Not Have Any Medical Treatment） at Treatment Day 84
Description: The patient was asked if she had any medical treatment (eg, prescribed medication, other treatment) because of her DUB during the past 12 weeks, and to specify the cost. The proportion of participants with such treatment are displayed.
Time Frame: Treatment day 84
Population: ITT, all participants with assessment at treatment day 84 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 119 | 65
Proportion of participants | 0.966 | 0.954

52. Secondary Outcome: Resource Use Assessment by Use of a Self Administered Questionnaire （Not Have Any Medical Treatment） at Treatment Day 196
Description: as for outcome 51
Time Frame: Treatment day 196
Population: ITT, all participants with assessment at treatment day 196 for this outcome measure
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 130 | 66
Proportion of participants | 0.977 | 0.985

53. Post Hoc Outcome: Proportion of Participants With Successful Treatment
Description: End of Study menstrual blood loss (MBL) ≤ 80 mL and a decrease to a value of ≤ 50% of the Baseline MBL was considered as treatment success.
Time Frame: during a time period of 28 days under treatment
Population: Only participants with heavy menstrual bleeding were included in the analysis.
Measure: Number; unit: Proportion of participants
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 132 | 75
Proportion of participants
  End of study MBL <=80 mL | 0.758 | 0.133
  Decrease MBL >=50% of baseline MBL | 0.788 | 0.133
  Successful treatment | 0.720 | 0.107

54. Post Hoc Outcome: Change in Absolute Value From Baseline Menstrual Blood Loss (MBL) to end-of Study MBL
Description: The MBL for each cycle includes intermenstrual bleeding in addition to withdrawal bleeding. Baseline MBL was the mean MBL of measured MBL during three cycles in the run-in Phase. One cycle was defined as 28 days. For this analysis, the run-in Phase was defined by the days 1 to 84 (= 3 cycles each of 28 days). End of Study MBL was measured during Cycle 7 of the Treatment Phase (data imputation and Last Observation Carried Forward was applied).
Time Frame: during a time period of 28 days under treatment
Population: Only participants with heavy menstrual bleeding were included in the analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Number analyzed (Participants) | 132 | 75
mL | -169.94 (225.762) | 4.628 (165.408)

ADVERSE EVENTS:
Arm/Group | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/145 | 2/81
Other Adverse Events (participants affected / at risk) | 44/145 | 21/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) (N=145) | Placebo (N=81)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Valerate/Dienogest (Natazia, Qlaira, BAY86-5027) (N=145) | Placebo (N=81)
Nasopharyngitis (Infections and infestations) | 12 (15) | 4 (4)
Serum ferritin decreased (Investigations) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 21 (46) | 12 (24)
Breast pain (Reproductive system and breast disorders) | 8 (10) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 8 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Schering AG is interested in the publication of the results of every study. As some of the information concerning the study drug and development activities at Schering AG may be of strictly confidential nature, any publication manuscript must first be reviewed by the sponsor before its submission or presentation.